CLINICAL TRIAL: NCT01654991
Title: A Randomized Trial of Home Versus Clinic-Based STD Testing Among Men
Brief Title: Randomized Trial of Home Versus Clinic-Based STD Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Peipert, Robert J. Terry Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201105031
Record Dates: First submitted 2012-07-29; First posted 2012-08-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Chlamydia; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinic-Based Testing (Active Comparator): Clinic-based STD screening using self-obtained urine samples in a local university clinical setting.
  Interventions: Behavioral: Clinic Screening
- Home-Based Testing (Experimental): Home-based STD screening using self-obtained urine samples and study paid postal return of samples.
  Interventions: Behavioral: Home Screening

INTERVENTIONS:
Behavioral: Home Screening — Home-based STD screening using self-obtained urine samples and study paid postal return of samples.
  Arms: Home-Based Testing
Behavioral: Clinic Screening — Clinic-based STD screening using self-obtained urine samples in a local university clinical setting.
  Arms: Clinic-Based Testing

SUMMARY:
This study randomizes St. Louis men to home-based STD screening or clinic-based STD screening. Home-based screening will be completed through the mail and clinic-based screening in a local clinical setting. We hypothesize that men randomized to home-based screening will be more likely to complete screening.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Ages 18-45
* Residing in St. Louis City or County
* English-speaking

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of men who complete testing in each study arm | 12 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Peipert, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Graseck AS, Secura GM, Allsworth JE, Madden T, Peipert JF. Home screening compared with clinic-based screening for sexually transmitted infections. Obstet Gynecol. 2010 Apr;115(4):745-752. doi: 10.1097/AOG.0b013e3181d4450d. PMID 20308834
- [Result] Graseck AS, Secura GM, Allsworth JE, Madden T, Peipert JF. Home compared with clinic-based screening for sexually transmitted infections: a randomized controlled trial. Obstet Gynecol. 2010 Dec;116(6):1311-1318. doi: 10.1097/AOG.0b013e3181fae60d. PMID 21099596
- [Result] Shih SL, Graseck AS, Secura GM, Peipert JF. Screening for sexually transmitted infections at home or in the clinic? Curr Opin Infect Dis. 2011 Feb;24(1):78-84. doi: 10.1097/QCO.0b013e32834204a8. PMID 21124216